CLINICAL TRIAL: NCT05135624
Title: SP16 as a Therapeutic for SARS-CoV-2 Induced ARDS
Brief Title: SP16 as a Therapeutic for COVID-19 Induced ARDS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial was terminated due to lack of patients.
Sponsor: Serpin Pharma, LLC (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRBHSR#210341
Record Dates: First submitted 2021-11-09; First posted 2021-11-26 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: SARS CoV 2 Infection; Pneumonia
Keywords: Pneumonia due to SARS-CoV-2
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Intervention Model Description: Cohort 1 - 7 subjects will be randomized to receive SP16 6 mg or placebo in a 7:3 ratio. Cohort 2 - 7 subject will be randomized to receive SP16 12 mg or placebo in a 7:3 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort dose 1 of SP16 (Experimental): Patients in cohort 1 (low dose SP16) will receive a single dose of SP16 (0.1 mg/kg or 6 mg) by subcutaneous injection
  Interventions: Drug: SP16 (6mg)
- Cohort dose 2 of SP16 (Experimental): Patients in cohort 2 (high dose SP16) will receive a single dose of SP16 (0.2 mg/kg or 12 mg) by subcutaneous injection
  Interventions: Drug: SP16 (12 mg)
- Placebo (Placebo Comparator): Patients in placebo arm will receive sterile water by subcutaneous injection.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SP16 (6mg) — SP16 will be administered as 2 concurrent, separate 2 mL s.c injections of 3mg/mL SP16
  Arms: Cohort dose 1 of SP16
Other: Placebo — Placebo will be administered as 2 concurrent, separate 2 mL s.c. injections of sterile water
  Arms: Placebo
Drug: SP16 (12 mg) — SP16 will be administered as a single 2 mL s.c. injection of 3 mg/mL SP16 and 1 concurrent separate 2 mL s.c. injection of sterile water
  Arms: Cohort dose 2 of SP16

SUMMARY:
This randomized, double-blind, placebo-controlled, Phase 1b study evaluates the safety and tolerability, and effects on cytokine and acute phase reactants of SP16, an anti-inflammatory drug, in patients with pneumonia due to SARS-CoV-2 infection. The study will enroll up to 20 patients and each eligible patient will be randomized to receive either one of two doses of SP16 (6 mg or 12 mg) or placebo by subcutaneous injection.

DETAILED DESCRIPTION:
SARS-CoV-2 infection is associated with excessive inflammation and cytokine storm that can result in lung damage and potentially severe disease. SP16 is an anti-inflammatory and homeostatic drug that rebalances innate immune responses potentially resulting in mitigation of inflammation and lung damage without immunosuppressive effects. SP16's mechanism of action is through targeting LRP1, a receptor that regulates a variety of physiological processes that contribute to inflammation and tissue injury, particularly in the lung. The main objective of this study is to determine the safety and tolerability, and effects on inflammation of SP16 administered subcutaneously at a dose of 6 mg (0.1 mg/kg) or 12 mg (0.2 mg/kg). SP16 has previously been well tolerated in both healthy individuals and heart attack patients at a dose of 0.2 mg/kg. The study will also evaluate improvements in clinical parameters such as patients requiring ventilation, improvement in blood oxygen levels (as defined by both SpO2 > 95% and respiratory rate ≤ 20/minute) and duration of hospitalization or time spent in the Intensive Care Unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible to participate in this study, the subject must meet all of the Inclusion criteria listed below:

* Hospitalized patients age ≥ 18 with diagnosis of SARS-CoV-2-infection based on positive
* PCR test result and can provide informed consent
* Diagnosed with pneumonia due to SARS-CoV-2
* Respiratory rate ≥ 25/minute and SpO2 ≤ 93%
* Review of Chest radiograph, chest computed tomography (CT) scan, or chest ultrasound consistent with bilateral infiltrates.
* Horowitz index (partial pressure of oxygen/fraction of inspired oxygen [PaO2/FiO2]) ≤ 300. If a subject does not have an arterial line in place, a SpO2/FiO2 ≤ 315 may be used.

Exclusion Criteria:

To be eligible for entry into the study, the subject must not meet any of the exclusion criteria listed below:

* Age < 18
* Pregnant or lactating women
* History of heart failure
* Clinically significant cardiac dysrhythmia, as determined by investigator
* History renal impairment
* Presence of any of the following abnormal laboratory values at screening: absolute neutrophil count (ANC) less than 2000 mm3, aspartate aminotransferase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of SP16 in subjects with pneumonia due to SARS-CoV-2 | Day 1 to 14
  Safety and tolerability of SP16 in subjects with pneumonia due to SARS-CoV-2 based on number of adverse events (AEs)
Change in inflammatory cytokines | Day 3, Day 6, and Day 14
  Subjects' change from baseline in plasma concentrations of inflammatory cytokines (IL-1β, TNF-α, IL-6, and IL-8)
Change in acute phase reactants | Day 3, Day 6, and Day 14
  Subjects' change from baseline of acute phase reactants (CRP, α-2 macroglobulin, fibrinogen, and D-dimer)

SECONDARY OUTCOMES:
Proportion of subjects requiring ventilation | Day 14
  The proportion of subjects in each dose group who required intubation and noninvasive ventilation by Day 14
Improvement from baseline in SpO2 | Days 3 and 14
  The proportion of subjects in each dose group who exhibited improvement from baseline in SpO2 levels, as defined by both SpO2 > 95% and respiratory rate ≤ 20/minute, at Days 3 and 14
Cumulative days on ventilator | Day 1 to 14
  Cumulative days on ventilator for each subject who required mechanical ventilation at any time during Day 1 to Day 14 period
Duration of hospitalization | Day 1 to 14
  Subjects' duration of hospitalization over the Day1 to Day 14 period
Time to clinical improvement | Day 1 to 14
  Subjects' time to clinical improvement (TTCI), which is defined as a National Early Warning Score 1 (NEWS2) of < 2 to be maintained for 24 h (during Days 1 to 14)
Proportion of subjects experiencing TTCI | Day 1 to 14
  The proportions of subjects in each cohort who experienced TTCI, which is defined as NEWS2 of < 2 to be maintained for 24 h
Subjects time to death | Day 1 to 14
  Subjects time to death or censoring over the period from Day 1 to Day 14 (subjects who withdraw prior to Day 14 will be censored on the day of withdrawal; subjects alive on Day 14 will be censored on Day 14)
Change from baseline in Horowitz index | Days 6 and 14
  Subjects' change from baseline on Days 6 and 14 in Horowitz index or in SpO2/FiO2
Subject's cumulative days in ICU | Day 1 to 14
  Subjects' cumulative number of days spent in the Intensive Care Unit (ICU) over Days 1 to 14

CONTACTS AND LOCATIONS:
Locations (1):
- UVA Health Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No